CLINICAL TRIAL: NCT00819260
Title: A Randomized Clinical Trial Comparing the Harmonic Scalpel to Electrocautery in Breast Reduction Surgery
Brief Title: Harmonic Scalpel Vs. Electrocautery in Breast Reduction Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant result achieved after enrollment of 31 of planned 50 subjects.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1182DF9
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Hyperplasia
Keywords: Mammaplasty; Electrocoagulation; Breast
MeSH Terms: conditions — Hyperplasia; Hyperthermia | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Harmonic Reduced Breast (Experimental): harmonic scalpel used to reduce breast on that side
  Interventions: Device: Harmonic Scalpel
- Electrocautery Reduced Breast (Active Comparator): Electrocautery (current practice = control) used to reduce breast on that side
  Interventions: Device: Electrocautery

INTERVENTIONS:
Device: Harmonic Scalpel — harmonic scalpel used to reduce breast on this side
  Arms: Harmonic Reduced Breast
Device: Electrocautery — Electrocautery used to reduce breast on this side
  Arms: Electrocautery Reduced Breast

SUMMARY:
Purpose: The aims of this randomized clinical trial are to assess and compare 3 different outcomes in women undergoing breast reduction surgery using two different surgical devices: the Harmonic Scalpel and electrocautery.

The three metrics are:

1. the time taken to complete the operation
2. drainage volume in the days immediately following surgery,
3. patient pain in the days immediately following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for enrollment if they agree to provide informed consent, can read and speak English, are at least 18 years of age, and are in generally good health.

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Kerrigan, MD, Principal Investigator — DHMC; Todd E Burdette, MD, Study Director — DHMC
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ran from January 2008 to January 2010. All patients were recruited in one surgical clinic at Dartmouth Hitchcock Medical Center.
Pre-assignment Details: Forty-three women were identified as potential study participants from May to December 2009. Three were excluded, because two were unable to consent and one was under 18 years old. Nine women declined to participate. Of the remaining 31 patients (72.1% of those identified), all completed the informed consent, the surgery, and the follow-up process.
Groups:
- All Participants: All participants were randomized to have one breast reduced using the harmonic scalpel and the other breast using electrocautery.
Period: Overall Study
Arm/Group | All Participants
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants randomized to have one breast reduced with harmonic scalpel and the other breast reduced with electrocautery.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age Continuous [Median (Full Range); unit: years] | 44 (0) [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Time for Operation
Description: Time to complete the breast reduction per breast.
Time Frame: day of surgery
Population: Women over the age of 18 who are not pregnant with symptomatic breast hypertrophy who underwent breast reduction surgery.
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | Harmonic Reduced Breast | Electrocautery Reduced Breast
Number analyzed (Participants) | 31 | 31
minutes | 32.9 (14.7) | 31 (8.1)

2. Secondary Outcome: Volume of Drainage in Surgical Drains
Description: An index was created to allow comparison between patients whose drain indwell times were different. This was created by taking total volume of drainage per breast drain and dividing it by the number of hours the drain was in place. The units are milliliters per hour.
Time Frame: within one week of surgery
Population: All participants in the study.
Measure: Median (Standard Deviation); unit: mL/hour
Arm/Group | Harmonic Reduced Breast | Electrocautery Reduced Breast
Number analyzed (Participants) | 31 | 31
mL/hour | 2.1 (1.4) | 2.8 (1.3)

3. Secondary Outcome: Pain Level in Surgical Sites
Description: An 11-point visual analog scale was used to obtain subjective pain levels from patients. 0 being no pain and 10 being worst pain imaginable.
Time Frame: first week after surgery
Population: all study participants
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Harmonic Reduced Breast | Electrocautery Reduced Breast
Number analyzed (Participants) | 31 | 31
units on a scale | 4 (3.2) | 4 (3)

4. Secondary Outcome: Hematoma
Description: A collection of blood or uncontrolled bleeding that necessitates a return to the operating room in the first day after surgery.
Time Frame: first day after surgery
Population: entire study population
Measure: Number; unit: participants
Arm/Group | Harmonic Reduced Breast | Electrocautery Reduced Breast
Number analyzed (Participants) | 31 | 31
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Harmonic Reduced Breast | Electrocautery Reduced Breast
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harmonic Reduced Breast (N=31) | Electrocautery Reduced Breast (N=31)
Infected seroma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Required operative evacuation, antibiotics and prolonged wound care.

LIMITATIONS AND CAVEATS:
We made a first analysis after 26 (intended enrollment 50) patients were enrolled and a result was strongly suggested. While the analysis was refined, 5 more patients enrolled. The study was then stopped after 31 patients enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No